CLINICAL TRIAL: NCT06498921
Title: Retrospective Observational Study With Nubeqa® (Darolutamide) for the Treatment of Adult Men With Metastatic Hormone Sensitive Prostate Cancer (mHSPC) in Combination With ADT and Docetaxel in BELGIUM
Brief Title: An Observational Study to Learn More About the Use of Darolutamide as a Part of a Combination Therapy in Belgian Men With Metastatic Hormone-Sensitive Prostate Cancer in Routine Medical Care
Acronym: BELBEQA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22743
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Hormone-sensitive Prostate Cancer
MeSH Terms: interventions — darolutamide; Androgen Antagonists; Docetaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- metastatic Hormone Sensitive Prostate Cancer (mHSPC): All adult men with a diagnosis of mHSPC, treated with darolutamide (Nubeqa, BAY1841788) in combination with androgen deprivation therapy (ADT) and docetaxel.
  Interventions: Other: Darolutamide (Nubeqa, BAY1841788) in combination with androgen deprivation therapy (ADT) and docetaxel

INTERVENTIONS:
Other: Darolutamide (Nubeqa, BAY1841788) in combination with androgen deprivation therapy (ADT) and docetaxel — No treatment will be provided to participants in the study. The decision on initiation of darolutamide (Nubeqa, BAY1841788) in combination with ADT and doctaxel and duration of treatment is solely at the discretion of the treating physician, guided by the recommendations outlined in the local product information.

SUMMARY:
This is an observational study in which only observations from routine clinical practices will be made. Participants will not receive any advice on treatment or any changes to healthcare as a part of the study.

In this study, medical records data of Belgian men with metastatic hormone sensitive prostate cancer (mHSPC) who had received or are receiving treatment with darolutamide in combination with androgen deprivation therapy (ADT) and docetaxel will be studied.

mHSPC is a cancer of the prostate gland, a male reproductive gland found below the bladder. Metastatic means that the cancer has spread to other parts of the body. Hormone-sensitive means it can be treated with hormone-therapy such as androgen deprivation therapy (ADT).

ADT lowers the level of androgens, male hormones, and slows down the growth of cancer cells. However, in some cases, ADT alone is not sufficient for the treatment of mHSPC and doctors recommend a combination of treatments.

The study drug darolutamide, in combination with ADT and docetaxel is an approved treatment for mHSPC. Darolutamide aims to work by blocking the androgens signals to slow the growth of the cancer cells. Docetaxel is a medicine used to treat different types of cancer and works by stopping the growth and spread of cancer cells.

The main purpose of this study is to learn more about the real-world use of darolutamide in combination with ADT and docetaxel in Belgian men with mHSPC.

To do this, researchers will study the following information about participants who are already prescribed this combination treatment by their treating doctors in real-word condition:

* Participants' cancer characteristics before starting the treatment, and
* Participants' treatment history The data will be collected between July 2024 to September 2024, from eligible participants' medical records.

Study doctors will only look at the medical records of adult men with mHSPC in Belgium.

In this study, only available data from routine care will be collected. No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with mHSPC
* Patients treated with darolutamide (Nubeqa, BAY1841788) in combination with ADT and docetaxel according to local reimbursement
* Initiation of treatment with darolutamide (Nubeqa, BAY1841788) in this indication between the index date (should be before 15MAR2024) and start of data collection.

Exclusion Criteria:

* Participation in an investigational program with interventions outside of routine clinical practice
* Contraindications according to the local reimbursement

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population of this study consists of all adult men with a diagnosis of mHSPC, treated with darolutamide (Nubeqa, BAY1841788) in combination with ADT and docetaxel, for this indication.
  mHSPC stands for metastatic Hormone Sensitive Prostate Cancer. ADT stands for androgen deprivation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Description of baseline characteristics of patients under real-word conditions | at baseline

SECONDARY OUTCOMES:
The average treatment duration with darolutamide (Nubeqa, BAY1841788) | up to 22 months
The therapeutic value of darolutamide (Nubeqa, BAY1841788) | up to 22 months

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Belgium

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.